CLINICAL TRIAL: NCT00801372
Title: Use of Existing Fibroblast Cells to Convert to Induced Pluripotent Stem Cells
Status: Recruiting | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Other Study IDs: 0522-08- HMO-CTIL
Record Dates: First submitted 2008-12-02; First posted 2008-12-03 (Estimated); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Pregnant, Healthy Females; Healthy Male Newborns
Keywords: termination of pregnancy; surgical circumcision; umbilical cord

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Existing bank of fibroblast cells retained.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pre-existing Fibroblast MCB: Pre-existing fibroblast donors for hESC derivation project

SUMMARY:
Induced pluripotent stem cells potentially may be useful in the future as an unlimited source of cells for transplantation.

The major goal of the project is to develop human iPS cells from existing lines of fibroblasts that were originally donated as clinical grade feeders for the development of clinical grade hESCs. The clinical grade feeders were developed from aborted fetuses, foreskin and umbilical cord.

DETAILED DESCRIPTION:
The potential to reprogram somatic cells into an embryonic state raises multiple basic research questions related both to the process of reprogramming and the properties of iPS cells. We will use various approaches to study the molecular mechanisms and processes that occur during reprogramming. We will use various experimental systems to characterize and study the properties of the iPS cells, their biology, developmental potential, capability to give rise to functional differentiated progeny etc.

The clinical grade donated feeders used in this project were developed under GMP conditions using animal-free reagents. For potential future clinical applications, the iPS cells will be developed under GMP conditions, using reagents and methods that will be acceptable for clinical applications.

ELIGIBILITY:
Inclusion Criteria:

* healthy, older than 18

Exclusion Criteria:

* non healthy, younger than 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: pregnant, healthy females older than 18 who signed an informed consent for the termination of the pregnancy.
  pregnant healthy couples older than 18 who signed an informed consent for a c-section.
  healthy male newborns, undergoing surgical circumcision who's parents older than 18 signed an informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2008-11 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin E Reubinoff, MD PhD, Principal Investigator — Chairman of Department of Obstetrics & Gynecology/IVF, Hadassah Ein Kerem
Locations (1):
- Hadassah Ein Kerem, Jerusalem, Israel, Israel

REFERENCES:
- [Background] Takahashi K, Tanabe K, Ohnuki M, Narita M, Ichisaka T, Tomoda K, Yamanaka S. Induction of pluripotent stem cells from adult human fibroblasts by defined factors. Cell. 2007 Nov 30;131(5):861-72. doi: 10.1016/j.cell.2007.11.019. PMID 18035408